CLINICAL TRIAL: NCT07292038
Title: A Phase I, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of NM6603 in Patients With Advanced Solid Tumors
Brief Title: Safety and Pharmacokinetics of NM6603 in Chinese Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NucMito Pharmaceuticals Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NM6603-CN-101
Record Dates: First submitted 2025-11-17; First posted 2025-12-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cancers
Keywords: advanced solid tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are enrolled in sequential dose-escalation cohorts using a traditional 3+3 design, in which each cohort receives an escalating dose of NM6603.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): NM6603, administered orally every day in 28-day cycles
  Interventions: Drug: NM6603

INTERVENTIONS:
Drug: NM6603 — NM6603 is an orally administered investigational small-molecule drug evaluated in this dose-escalation study in patients with advanced solid tumors.

SUMMARY:
This study is to assess the MTD and PK of NM6603 in adult patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1, open label, 3+3 dose escalation study designed to evaluate the safety profile, the maximum tolerated dose (MTD), the pharmacokinetic and the preliminary antitumor activity of NM6603 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors (primarily advanced colorectal cancer or triple-negative breast cancer) confirmed by histology or cytology
* Prior adequate standard therapy with documented progression or intolerance, or lack of available standard therapy options, or contraindications to standard therapy
* At least one evaluable tumor lesion per RECIST version 1.1
* Age 18 to 75 years at the time of informed consent
* Body weight 45 kg or greater for men and 40 kg or greater for women
* ECOG performance status 0 or 1
* Expected survival time greater than 12 weeks
* Adequate organ and bone marrow function as defined below:

  * Absolute neutrophil count 1500 per mm3 or greater
  * Platelet count 100000 per mm3 or greater with no transfusion or growth factor use within 14 days before first dose
  * Hemoglobin 9.0 g/dL or greater with no transfusion or stimulating factors within 14 days before first dose
  * Total bilirubin 1.5 times upper limit of normal (ULN) or less (patients with Gilbert syndrome allowed)
  * AST and ALT 2.5 times ULN or less without liver metastasis, or 5 times ULN or less with liver metastasis
  * Creatinine clearance 60 mL/min or greater (Cockcroft-Gault formula)
  * INR 1.5 times ULN or less and APTT 1.5 times ULN or less
* Male subjects and female subjects of childbearing potential agree to use effective contraception from signing consent until 6 months after last dose; men must not donate sperm; women of childbearing potential require a negative pregnancy test within 7 days prior to first dose
* Able and willing to comply with study visits, procedures, and provide written informed consent

Exclusion Criteria:

* Known hypersensitivity to NM6603 or its components
* Prior treatment with a drug targeting the same mechanism of action or molecular target
* Participation in another drug or device clinical trial within 4 weeks before first dose
* Major surgery within 4 weeks before first dose or planned surgery during the study
* Chemotherapy, biologic therapy, macromolecular targeted therapy, or radiotherapy within 4 weeks before first dose
* Oral fluoropyrimidines or other small molecule targeted agents received within 2 weeks or 5 half-lives before first dose (whichever is longer)
* Use of traditional Chinese medicine or herbal products with antitumor activity within 2 weeks before first dose
* Use of medications known to prolong QT interval or strong inhibitors or inducers of CYP1A2, CYP2A6, or CYP3A4 within 7 days before first dose, or requirement for continued use
* Systemic corticosteroids or immunosuppressive drugs at doses greater than 10 mg/day prednisone or equivalent within 4 weeks before first dose (physiologic replacement and topical/inhaled forms allowed)
* History of another malignancy within 5 years except for curatively treated carcinoma in situ of the cervix, non-melanoma skin cancer, localized prostate cancer, or ductal carcinoma in situ
* Active central nervous system metastases, including symptomatic brain metastases, leptomeningeal disease, spinal cord compression, or unstable brain metastasis
* Treated brain metastases allowed if stable for 4 weeks or longer, no neurologic symptoms, and not receiving systemic corticosteroids above replacement dose for 4 weeks
* Untreated asymptomatic brain metastases 1.5 cm or smaller allowed if not requiring corticosteroids
* Uncontrolled disease including:

  * Active infection
  * Acute coronary syndrome, symptomatic heart failure (NYHA class 2 or greater), cerebrovascular accident, transient ischemic attack, stroke, deep vein thrombosis, pulmonary embolism, aneurysm, arterial dissection, or other grade 3 or higher cardiovascular or cerebrovascular events within 6 months
  * Left ventricular ejection fraction less than 50 percent, uncontrolled hypertension (systolic over 160 mmHg or diastolic over 100 mmHg), uncontrolled hyperglycemia, ventricular arrhythmias requiring intervention, second or third degree AV block, congenital long QT syndrome, QTcF greater than 450 ms
  * Active peptic ulcer, gastritis, or bleeding disorder
  * Risk factors for pancreatitis including history of pancreatitis, uncontrolled hyperlipidemia, excessive alcohol use, uncontrolled diabetes, gallbladder disease, or medications associated with elevated triglycerides or pancreatic toxicity
  * Psychiatric or social conditions that may affect study compliance or ability to provide informed consent
* Family history of long QT syndrome or unexplained sudden death before age 40 in a first-degree relative
* Inability to swallow oral medication or gastrointestinal disease or major GI surgery likely to impair drug absorption, metabolism, or excretion
* Known alcohol or substance dependence
* Active syphilis; positive HIV antibody; positive HCV antibody with detectable HCV RNA; active hepatitis B infection (HBsAg positive with HBV DNA 1000 IU/mL or greater)
* Not recovered to grade 1 or less from prior therapy toxicity (NCI CTCAE v5.0), except for alopecia, irreversible grade 1 fatigue, or clinically insignificant lab abnormalities such as lymphocyte count decrease
* Pregnant or breastfeeding women or women planning pregnancy during the study
* Any condition that, in the investigator's judgment, makes the subject unsuitable or may affect compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | During the first cycle. Each cycle is 28 days
  MTD was defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients. DLT will be defined as toxicities that meet pre-defined severity criteria(according to the NCI CTCAE v5.0 toxicity assessment criteria), and assessed as having a suspected relationship to study drug that occurred within the first cycle(28 days) of treatment.
Recommended Phase II Dose | Up to 1 Year
  The recommended dosage for subsequent Phase II studies will be based on MTD (Maximum Tolerant Dose), pharmacokinetics, preliminary efficacy and safety data from the study

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of NM6603 | Up to 31 days
  To evaluate the maximum observed concentration (Cmax) of NM6603 in subjects with advanced solid tumors
Time of maximum observed concentration (Tmax) of NM6603 | Up to 31 days
  To evaluate the time of maximum observed concentration (Tmax) of NM6603 in subjects with advanced solid tumors
Terminal elimination half-life (t1/2) of NM6603 | Up to 31 days
  To evaluate the terminal elimination half-life (t1/2) of NM6603 in subjects with advanced solid tumors
Area under the curve from the time of dosing to the time of the last measurable concentration (AUClast) of NM6603 | Up to 31 days
  To evaluate the area under the curve from the time of dosing to the time of the last measurable concentration (AUClast) of NM6603 in subjects with advanced solid tumors
Area under the curve from the time of dosing to infinity (AUCinf) of NM6603 | Up to 31 days
  To evaluate the area under the curve from the time of dosing to infinity (AUCinf) of NM6603 in subjects with advanced solid tumors
Efficacy of NM6603 by Overall response rates (ORR) | Up to 1 year
  Overall response rate (ORR) defined as the proportion of participants with complete response (CR) or partial response (PR) as determined by the investigator using RECIST V1.1.
Efficacy of NM6603 by disease control rate (DCR) | Up to 1 year
  Disease control rate (DCR) is defined as the percentage of subjects who achieve complete response, partial response, or stable disease according to RECIST version 1.1.
Efficacy of NM6603 by Overall Survival (OS) | Up to a year
  Overall survival is defined as the time from the first dose of study treatment until death from any cause.
Safety of NM6603 by incidence and severity of treatment-emergent adverse events (TEAEs) | Up to 1 year
  The number of subjects experiencing treatment-emergent adverse events will be recorded, and the severity of each event will be graded according to NCI CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University Cancer Center (SYSUCC), Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No